CLINICAL TRIAL: NCT06304623
Title: The Role of Cellular Therapy With SVF Cells (Stromal Vascular Fraction) of Adipose Tissue Origin in the Treatment of Pulmonary Fibrosis Post COVD-19
Brief Title: SVF for Treating Pulmonary Fibrosis Post COVID-19
Acronym: SVFCOVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael H Carstens (Other)
Collaborators: Ministerio de Salud de Nicaragua (Unknown); Wake Forest University (Other); National Autonomous University of Nicaragua (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRE.112
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SVF cells treatment (Experimental): 40 subjects were treated with autologous SVF intravenous treatment.
  Interventions: Biological: Autologous adipose-derived SVF IV administration

INTERVENTIONS:
Biological: Autologous adipose-derived SVF IV administration — Subjects received an intravenous injection of autologous adipose-derived SVF.

SUMMARY:
General description of the study

This is a prospective, multicenter, expanded access interventional study of subjects recovered from COVID-19 pneumonia to assess their response to intravenous administration of adipose-derived autologous SVF.

Primary objective

The purpose of this study was to evaluate the safety of single intravenous injections of autologous adipose-derived SVF produced using the GID SVF-2 device system for the treatment of secondary respiratory distress associated with COVID-19.

Secondary objective

To evaluate the efficacy of the initial treatment with SVF IV.

DETAILED DESCRIPTION:
The recent outbreak of Coronavirus 2 (SARS-CoV-2) has spread rapidly throughout the world, resulting in a global pandemic with devastating socioeconomic consequences. After being declared a public health emergency by the World Health Organization (WHO), there is an urgent need to develop effective therapeutic strategies for critically ill COVID-19 patients. This new virus strain causes a complex disease with a wide range of presentations, from mild symptoms to multi-organ failure. A common feature of severe cases is the pathologically complex "cytokine storm" that presents as an excessive immune response with rapid progression of disease and high mortality. In particular, the severe outcomes of SARS CoV-2 are associated with elevated C-reactive protein and Interleukin-6 in the lungs. COVID-19 infection can rapidly decompensate into severe respiratory failure requiring intubation and mechanical ventilation. The need for mechanical ventilation portends a poor prognosis, with a reported mortality rate of up to 88%.

Survivors of COVID-19 pneumonia face sequelae of their disease that affect multiple organ systems. In particular, a significant number present with ongoing problems of breathlessness and reduced oxygenation, turning previously healthy patients into virus-induced pulmonary cripples. The mechanism for this is the intense scarring and destruction of the microcirculation found in the lungs of COVID-19 survivors. There is an urgent need for the development of treatment protocols that are capable of reducing the degree of pulmonary fibrosis and promoting local angiogenesis to better support injured alveoli.

In recent decades, mesenchymal stromal cells (MSCs) have emerged as a potential therapeutic agent for cell-based therapies due to the beneficial effects on immunomodulation and tissue repair/regeneration. These cells possess properties unique self-renewal and capacity to differentiate into multiple lineages. MSCs are found in small numbers in bone marrow (BMSC) and umbilical cord tissue. MSCs are also found in adipose tissue (referred to as ASCs) where they exist as part of a multicellular population, the stromal vascular fraction (SVF). ASC populations are 500-1000 more abundant than their bone marrow counterparts.

Adipose tissue provides a source of Stromal Vascular Fraction (SVF) that can be isolated and transplanted to the patient during the same surgical procedure, at the point of care. SVF is a heterogeneous mixture of stromal progenitor cells, pericytes, endothelial precursor cells, and macrophages. Acting collectively, SVF has been shown to possess broad anti-inflammatory and regenerative properties. SVF has been shown to be safe after IV administration and has shown some promising results in restoring respiratory function in patients with severe lung disorders. Based on public analysis of single cell RNA sequencing (scRNA-seq) data, SVF demonstrates the absence of ACE2 expression, indicating its potential as a resistant phenotype to SARS-CoV-2 infection. In Taken together, IV administration of adipose- derived SVF is presented as a novel treatment approach to improve the clinical outcome of respiratory-compromised COVID-19 patients.

The clinical impact of SVF for COVID-19 is based on 5 mechanisms of action. These have been widely documented (see attached publications and bibliography).

Anti-inflammatory Immunomodulation, especially T-regs Antifibrosis. Matrix metalloproteinases and liver growth factor. Support for regenerative cell populations in situ. Lung asthma studies Angiogenesis under ischemic conditions, based on the release of VEGF.

Therapy with SVF cells from adipose tissue is advantageous as large numbers of cells can be removed from small volumes (30-90 cc) by a minimally invasive liposuction procedure.

Indication for expanded access

This is an expanded access study to treat a small group of subjects with pulmonary sequelae after recovery from COVID-19 pneumonia of autologous adipose-derived SVF administered using as single intravenous injection.

Objectives of clinical research

Main objective

To assess the safety of a single injection of autologous adipose-derived SVF produced with the GID SVF-2 device for the treatment of respiratory distress.

associated with COVID-19.

Secondary objective

To assess efficacy, by (1) maintaining SaO2 saturation ≥ at the existing level on noninvasive oxygen support, (2) achieving a reduction in the level of oxygen support required to maintain SaO2 ≥ 92, using intravenous injection of autologous adipose derived SVF produced using the GID SVF-2 device system for the treatment of respiratory distress associated with COVID-19.

Expected duration of the clinical investigation

Follow-up controls at 3, 6, 9, and 12 months. The total duration of the study is 1 year.

Clinical Protocol

Study design

General study design

This is a prospective, multicenter, expanded access interventional study of subjects with COVID-19. Forty (40) subjects with confirmed COVID-19 and SaO2 ≤ 92 were treated. Subjects received an intravenous injection of autologous adipose-derived SVF. Subjects will be followed for 6 weeks.

Study procedures

Detection procedures

The initial evaluation was done at the local Centro de Salud. Subjects were then referred to HEODRA or HECAM for confirmatory diagnosis and additional tests.

Concomitant medications

All concomitant medications considered Standard of Care are accepted. A concomitant medication case report form will be completed at each subject follow-up visit.

Summary of study treatment

40 non-randomized patients will be treated with autologous SVF. Minimum dosage: 45x106 ± 5x106 cells Treatment plan: a single intervention

Follow-up Serum samples (20 cc) - inflammation factors: 1 month, 3 months, 6 months PFTs + DLco: preop, 1 month, 3 months, 6 months weeks, and 12 months CT: preop, 3 months, 6 months, 12 months SF-36 quality of life questionnaire SF-36 (Medical Outcomes Trust): pre-op, 12 months SGRQ-C respiratory questionnaire SGRQ-C (St. George's University): pre-op, 12 months

The subject's adipose tissue will be acquired by liposuction of the abdomen or flanks and placed directly into the GID SVF-2 device. The harvested adipose tissue will be enzymatically digested in the same GID SVF-2 device using the GIDZyme-2-70 enzyme and centrifuged in the same GID SVF-2 device to concentrate the SVF cells. SVF cells will be removed and an active treatment dose of 45 x 106 (±5 x 106) SVF cells will be injected into a 100 ml IV bag containing LR. Fluids will be given through an IV catheter through a blood filter over 10 minutes.

Dosage

Dose preparation

Using the LunaStem® Nucleocounter Cell Concentration and Dilution Factor 100 calculate the volume needed using the following equation and transfer that amount of resuspension to a 10 mL syringe.

#ml = dose = 40 x 106 (+/- 5x106)

Dose administration The way to administer SVF for vascular use is the same whether it is intravenous (IV) or intravenous (IA).

The treatment was administered intravenously using an intravenous catheter with a blood filter.

Add the dose to a 100 ml bag of LR that has been warmed to 37°C and mix well. Administer the 100 ml over 10 minutes.

Adherence to treatment

Each subject had time to read the consent form and ask questions about the study before signing the informed consent. Subjects should contact the physician or staff if participant have any concerns during the study. It will be emphasized that the subject must comply with the protocol and be honest about her symptoms.

Withdrawal of subjects for non-compliance

Subjects may be terminated from the study at the discretion of the principal investigator only for reasons related to study examinations that would jeopardize the subject's health and/or welfare if participants were to continue in the study. Subjects may voluntarily withdraw from the study at any time without prejudice.

• Subjects withdrawn will not be replaced if participant have received study treatment.

Schedule of study visits

The initial evaluation and informed consent took place in the hospitals. Prior to treatment, subjects were evaluated to determine if participant meet the inclusion/exclusion criteria. If not already provided, demographics, medical history, concomitant medications, SaO2, and arterial blood gases was collected. The subject were enrolled if participant meet all the eligibility criteria and have signed the Informed Consent.

The time between enrollment and treatment not exceeded 48 hours.

On the day of treatment, each subject was reassessed for inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

Patients were identified at Managua and Leon, Nicaragua, community health centers and screened for eligibility by study physicians.

* Forty PCR-confirmed COVID-19 patients
* Persistent pulmonary complaints of dyspnea for at least 2 months after hospital discharge.
* Age 18 - 85 years.
* Male or Female.
* A body mass index of > 22.
* Forced vital capacity (FVC) > 40% predicted and < 70% predicted
* Diffusing lung capacity of the lungs for carbon monoxide (DLCO) > 20% predicted and < 70% predicted.

Exclusion Criteria:

* Use of home oxygen
* History of pulmonary malignancy.
* Immunosuppressive drug treatment
* History of prior cardiac disease with an ejection fraction of ≤30%
* Diabetes
* Pregnancy or plans to conceive during the study period.
* Participation in another clinical study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Safety of treatment with SVF IV | Up to 12 months post injection.
  None of the participants with potential pulmonary severe adverse events (SAE) related to the SVF cell infusion of single intravenous injection of autologous adipose-derived SVF produced using the GID SVF-2 device system.

SECONDARY OUTCOMES:
Efficacy of the initial treatment with SVF IV | Up to 12 months
  All subjects with Dyspnea symptoms improved: Mechanical function of the lung by spirometry increased in forced vital capacity (FVC).

OTHER OUTCOMES:
Effectiveness of the initial treatment with SVF IV | Up to 12 months
  All subjects with Alveolar-capillary diffusion of oxygen enhanced using the diffusing capacity of the lung for carbon monoxide (DLCO) metric.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Lopez, MD, Study Director — Hospital Escuela Oscar Danilo Rosales, Leon (HEODRA); Yanury Dolmus, MD, Study Director — Hospital Escuela Cesar Amador Molina, Matagalpa (HECAM)
Locations (2):
- Nicaragua (2):
  - Hospital Escuela Oscar Danilo Rosales Arguello (HEODRA), León, León Department
  - Hospital Escuela Cesar Amador Molina, Matagalpa

REFERENCES:
- [Background] Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species Severe acute respiratory syndrome-related coronavirus: classifying 2019-nCoV and naming it SARS-CoV-2. Nat Microbiol. 2020 Apr;5(4):536-544. doi: 10.1038/s41564-020-0695-z. Epub 2020 Mar 2. PMID 32123347
- [Background] WHO Director-General's opening remarks at the media briefing on COVID-19 - 11 March2020. https://www.who.int/dg/speeches/detail/who-director-general-s-opening-remarks-at-the- media-briefing-on-covid-19---11-march-2020. Published 2020
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Jiang S, Du L, Shi Z. An emerging coronavirus causing pneumonia outbreak in Wuhan, China: calling for developing therapeutic and prophylactic strategies. Emerg Microbes Infect. 2020 Jan 31;9(1):275-277. doi: 10.1080/22221751.2020.1723441. eCollection 2020. No abstract available. PMID 32005086
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Weiss P, Murdoch DR. Clinical course and mortality risk of severe COVID-19. Lancet. 2020 Mar 28;395(10229):1014-1015. doi: 10.1016/S0140-6736(20)30633-4. Epub 2020 Mar 17. No abstract available. PMID 32197108
- [Background] Pittenger MF, Discher DE, Peault BM, Phinney DG, Hare JM, Caplan AI. Mesenchymal stem cell perspective: cell biology to clinical progress. NPJ Regen Med. 2019 Dec 2;4:22. doi: 10.1038/s41536-019-0083-6. eCollection 2019. PMID 31815001
- [Background] Nauta AJ, Fibbe WE. Immunomodulatory properties of mesenchymal stromal cells. Blood. 2007 Nov 15;110(10):3499-506. doi: 10.1182/blood-2007-02-069716. Epub 2007 Jul 30. PMID 17664353
- [Background] Le Blanc K, Davies LC. Mesenchymal stromal cells and the innate immune response. Immunol Lett. 2015 Dec;168(2):140-6. doi: 10.1016/j.imlet.2015.05.004. Epub 2015 May 15. PMID 25982165
- [Background] Chamberlain G, Fox J, Ashton B, Middleton J. Concise review: mesenchymal stem cells: their phenotype, differentiation capacity, immunological features, and potential for homing. Stem Cells. 2007 Nov;25(11):2739-49. doi: 10.1634/stemcells.2007-0197. Epub 2007 Jul 26. PMID 17656645
- [Background] Nguyen A, Guo J, Banyard DA, Fadavi D, Toranto JD, Wirth GA, Paydar KZ, Evans GR, Widgerow AD. Stromal vascular fraction: A regenerative reality? Part 1: Current concepts and review of the literature. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):170-9. doi: 10.1016/j.bjps.2015.10.015. Epub 2015 Oct 31. PMID 26565755
- [Background] Brown, P, Katz AJ. Adipose -derived stem cells In: Atala A (ed). Textbook of Regenerative Medicine Elsevier, 3rd ed. 2019, pp.
- [Background] Kapur SK, Dos-Anjos Vilaboa S, Llull R, Katz AJ. Adipose tissue and stem/progenitor cells: discovery and development. Clin Plast Surg. 2015 Apr;42(2):155-67. doi: 10.1016/j.cps.2014.12.010. PMID 25827560
- [Background] Guo J, Nguyen A, Banyard DA, Fadavi D, Toranto JD, Wirth GA, Paydar KZ, Evans GR, Widgerow AD. Stromal vascular fraction: A regenerative reality? Part 2: Mechanisms of regenerative action. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):180-8. doi: 10.1016/j.bjps.2015.10.014. Epub 2015 Oct 24. PMID 26546112
- [Background] Regmi S, Pathak S, Kim JO, Yong CS, Jeong JH. Mesenchymal stem cell therapy for the treatment of inflammatory diseases: Challenges, opportunities, and future perspectives. Eur J Cell Biol. 2019 Dec;98(5-8):151041. doi: 10.1016/j.ejcb.2019.04.002. Epub 2019 Apr 14. PMID 31023504
- [Background] Limper AH. Safety of IV Human Mesenchymal Stem Cells in Patients With Idiopathic Pulmonary Fibrosis. Chest. 2017 May;151(5):951-952. doi: 10.1016/j.chest.2016.12.015. No abstract available. PMID 28483127
- [Background] Comella K, Blas JAP, Ichim T, Lopez J, Limon J, Moreno RC. Autologous Stromal Vascular Fraction in the Intravenous Treatment of End-Stage Chronic Obstructive Pulmonary Disease: A Phase I Trial of Safety and Tolerability. J Clin Med Res. 2017 Aug;9(8):701-708. doi: 10.14740/jocmr3072w. Epub 2017 Jul 1. PMID 28725319
- [Background] Michalek J, Vrablikova A, Heinrich KG, Dudasova Z. Stromal Vascular Fraction Cell Therapy for a Stroke Patient-Cure without Side Effects. Brain Sci. 2019 Mar 6;9(3):55. doi: 10.3390/brainsci9030055. PMID 30845656
- [Background] Turner AJ, Hiscox JA, Hooper NM. ACE2: from vasopeptidase to SARS virus receptor. Trends Pharmacol Sci. 2004 Jun;25(6):291-4. doi: 10.1016/j.tips.2004.04.001. PMID 15165741
- [Background] Leng Z, Zhu R, Hou W, Feng Y, Yang Y, Han Q, Shan G, Meng F, Du D, Wang S, Fan J, Wang W, Deng L, Shi H, Li H, Hu Z, Zhang F, Gao J, Liu H, Li X, Zhao Y, Yin K, He X, Gao Z, Wang Y, Yang B, Jin R, Stambler I, Lim LW, Su H, Moskalev A, Cano A, Chakrabarti S, Min KJ, Ellison-Hughes G, Caruso C, Jin K, Zhao RC. Transplantation of ACE2- Mesenchymal Stem Cells Improves the Outcome of Patients with COVID-19 Pneumonia. Aging Dis. 2020 Mar 9;11(2):216-228. doi: 10.14336/AD.2020.0228. eCollection 2020 Apr. PMID 32257537
- [Background] Caplan AI, Correa D. The MSC: an injury drugstore. Cell Stem Cell. 2011 Jul 8;9(1):11-5. doi: 10.1016/j.stem.2011.06.008. PMID 21726829
- [Background] Gutta S, Grobe N, Kumbaji M, Osman H, Saklayen M, Li G, Elased KM. Increased urinary angiotensin converting enzyme 2 and neprilysin in patients with type 2 diabetes. Am J Physiol Renal Physiol. 2018 Aug 1;315(2):F263-F274. doi: 10.1152/ajprenal.00565.2017. Epub 2018 Mar 21. PMID 29561187
- [Background] Giannandrea M, Parks WC. Diverse functions of matrix metalloproteinases during fibrosis. Dis Model Mech. 2014 Feb;7(2):193-203. doi: 10.1242/dmm.012062. PMID 24713275
- [Background] Pardo A, Cabrera S, Maldonado M, Selman M. Role of matrix metalloproteinases in the pathogenesis of idiopathic pulmonary fibrosis. Respir Res. 2016 Mar 4;17:23. doi: 10.1186/s12931-016-0343-6. PMID 26944412
- [Background] Crestani B, Marchand-Adam S, Quesnel C, Plantier L, Borensztajn K, Marchal J, Mailleux A, Soler P, Dehoux M. Hepatocyte growth factor and lung fibrosis. Proc Am Thorac Soc. 2012 Jul;9(3):158-63. doi: 10.1513/pats.201202-018AW. PMID 22802291
- [Background] Castro LL, Kitoko JZ, Xisto DG, Olsen PC, Guedes HLM, Morales MM, Lopes-Pacheco M, Cruz FF, Rocco PRM. Multiple doses of adipose tissue-derived mesenchymal stromal cells induce immunosuppression in experimental asthma. Stem Cells Transl Med. 2020 Feb;9(2):250-260. doi: 10.1002/sctm.19-0120. Epub 2019 Nov 20. PMID 31746562
- [Background] Zakhari JS, Zabonick J, Gettler B, Williams SK. Vasculogenic and angiogenic potential of adipose stromal vascular fraction cell populations in vitro. In Vitro Cell Dev Biol Anim. 2018 Jan;54(1):32-40. doi: 10.1007/s11626-017-0213-7. Epub 2017 Dec 1. PMID 29197029
- [Background] Carstens MH, Gomez A, Cortes R, Turner E, Perez C, Ocon M, Correa D. Non-reconstructable peripheral vascular disease of the lower extremity in ten patients treated with adipose-derived stromal vascular fraction cells. Stem Cell Res. 2017 Jan;18:14-21. doi: 10.1016/j.scr.2016.12.001. Epub 2016 Dec 8. PMID 27984756